CLINICAL TRIAL: NCT02475369
Title: Pilot Study of the Efficacy of Pancreatic Enzyme Supplementation for Symptom Control in Celiac Disease Not Responding to the Gluten Free Diet
Brief Title: Pancreatic Enzyme Supplementation for Celiac Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial was terminated prematurely by the sponsor for administrative reasons.
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Actavis Inc. (Industry)
Responsible Party: Principal Investigator, Ciaran Kelly, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2014P000375
Record Dates: First submitted 2015-06-16; First posted 2015-06-18 (Estimated); Results first posted 2021-02-08 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-04

CONDITIONS: Celiac Disease
Keywords: pancreatic enzyme supplementation
MeSH Terms: conditions — Celiac Disease | interventions — Pancrelipase; Lipase; Peptide Hydrolases; Amylases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PES, Then Placebo (Other): Participants first received Pancreatic Enzyme Supplementation (PES) for 10 days. PES taken 6 times daily with gluten free meals and snacks. To facilitate duodenal digestion Omeprazole (20 mg/QD) was co-administered. After a washout period of 1 week, they then received placebo tablets (matching PES treatment) 6 times daily for 10 days.
  Interventions: Drug: pancrelipase
- Placebo, Then PES (Other): Participants first received placebo tablets (matching PES) for 10 days. Placebo was taken 6 times daily with gluten-free meals and snacks. To facilitate duodenal digestion Omeprazole (20 mg/QD) was co-administered. After a washout period of 1 week, they then received PES tablets six times daily for 10 days.
  Interventions: Drug: pancrelipase

INTERVENTIONS:
Drug: pancrelipase
  Other Names: Viokase; lipase, protease, amylase

SUMMARY:
The purpose of this protocol is to conduct a pilot study to investigate whether pancreatic enzyme supplementation will improve symptoms in individuals with celiac disease who suffer persistent symptoms despite a gluten free diet. This protocol specifically aims to:

1. Evaluate the efficacy of pancreatic enzyme supplementation for reduction of gastrointestinal symptoms in patients with celiac disease on a gluten free diet.
2. Assess the ability of fecal elastase levels to predict response to pancreatic enzyme supplementation in patients with celiac disease on a gluten free diet.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven celiac disease.
* Age 18-80.
* Ongoing symptoms defined as a CeD-GSRS score of greater than 3 during the run in period.
* Subject must be following a gluten free diet.
* tTG < 40 units at screening.

Exclusion Criteria:

* Taking prescription or over the counter enzyme supplements for 1 month prior to enrollment.
* Pregnant, breastfeeding or planning pregnancy. Woman using acceptable methods of contraception will be included. Acceptable methods of contraception include oral hormonal contraceptives, implanted hormonal contraceptives, diaphragm with spermicide, condoms, intra-uterine device, abstinence, and male partner vasectomy.
* Patients with a pork allergy or who are unwilling to consume pork products.
* English proficiency unsuitable for completion of surveys.
* Known severe pancreatic disease.
* Known history of prior cancer (except squamous or basal cell skin cancer).
* Patients with lactose intolerance who are unable to tolerate a minimum of 1oz (2 tablespoons) of whole milk per day.
* Clinically significant abnormality in safety lab values (i.e. CBC and BMP) at screening that may impact subject safety or the scientific integrity of the study.
* Other known active GI condition including but not limited to inflammatory bowel disease, small intestine bacterial overgrowth, and obvious FODMAP intolerance.
* History of all major gastrointestinal surgery other than appendectomy or cholecystectomy.
* Comorbid condition that in the opinion of the investigator would interfere with the subject's participation in the study or would confound the results of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-05; Primary Completion 2019-06 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ciaran Kelly, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Kelly CP, Green PH, Murray JA, Dimarino A, Colatrella A, Leffler DA, Alexander T, Arsenescu R, Leon F, Jiang JG, Arterburn LA, Paterson BM, Fedorak RN; Larazotide Acetate Celiac Disease Study Group. Larazotide acetate in patients with coeliac disease undergoing a gluten challenge: a randomised placebo-controlled study. Aliment Pharmacol Ther. 2013 Jan;37(2):252-62. doi: 10.1111/apt.12147. Epub 2012 Nov 19. PMID 23163616
- [Background] Svedlund J, Sjodin I, Dotevall G. GSRS--a clinical rating scale for gastrointestinal symptoms in patients with irritable bowel syndrome and peptic ulcer disease. Dig Dis Sci. 1988 Feb;33(2):129-34. doi: 10.1007/BF01535722. PMID 3123181
- [Derived] Yoosuf S, Barrett CG, Papamichael K, Madoff SE, Kurada S, Hansen J, Silvester JA, Therrien A, Singh P, Dennis M, Leffler DA, Kelly CP. Pancreatic enzyme supplementation versus placebo for improvement of gastrointestinal symptoms in non-responsive celiac disease: A cross-over randomized controlled trial. Front Med (Lausanne). 2023 Jan 4;9:1001879. doi: 10.3389/fmed.2022.1001879. eCollection 2022. PMID 36687454

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for eligibility between 4/16/2015 and 5/28/2017 at Beth Israel Deaconess Medical Center in Boston Massachusetts
Pre-assignment Details: 21 participants were randomized.
Period: Run-in Washout Period #1 (7 Days)
Arm/Group | PES, Then Placebo | Placebo, Then PES
Started | 10 | 11
Completed | 3 | 9
Not Completed | 7 | 2
Not completed — Sponsor terminated study prematurely | 7 | 2
Period: Treatment Period #1 (10 Days)
Arm/Group | PES, Then Placebo | Placebo, Then PES
Started | 3 | 9
Completed | 3 | 9
Not Completed | 0 | 0
Period: Run-in Washout Period #2 (7 Days)
Arm/Group | PES, Then Placebo | Placebo, Then PES
Started | 3 | 9
Completed | 3 | 9
Not Completed | 0 | 0
Period: Treatment Period #2 (10 Days)
Arm/Group | PES, Then Placebo | Placebo, Then PES
Started | 3 | 9
Completed | 3 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Treatments: The treatment phase was comprised of two 10-day treatment periods. The study began with a 7 day washout period followed by Treatment period 1. After 10 day treatment period one all participants received a 7 day washout run-in period. Finally, all patients received a 10 day treatment period 2. Participants were randomized to two groups which were "PES, then Placebo" (n=3) or "Placebo, then PES" (n=9). Per cross-over design, all subjects have received both intervention at the end of the trial.
Arm/Group | All Study Treatments
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 42 [24 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Baseline Celiac Disease Gastrointestinal Symptom (CeD-GSRS)Response Scale [Median (Full Range); unit: units on a scale] — Celiac Disease Gastrointestinal Symptom Response Scale:scores range from 1 to 7, with greater scores indicating worse symptoms. The minimum score obtainable is 15 and the maximum score obtainable is 105. This is then divided by 15 to obtain the minimum overall CeD-GSRS score of 1 and maximum of 7. It has 3 domains- Abdominal pain, Indigestion and Diarrhea domains, each domain having a score ranging from 1-7. The higher the overall score, the more severe the symptoms.
  units on a scale | 3.25 [2.30 to 4.30]
Baseline Celiac Symptom Index (CSI) [Median (Full Range); unit: units on a scale] — Celiac Symptom Index: scores range from 16 to 80, with greater scores indicating worse symptoms
  units on a scale | 35 [26 to 57]
Baseline abdominal pain on Celiac Disease Gastrointestinal Symptom Response Scale (CeD-GSRS) [Median (Full Range); unit: units on a scale] — Celiac Disease Gastrointestinal Symptom Response Scale:scores range from 1 to 7, with greater scores indicating worse symptoms. On the domain of abdominal pain the minimum score is 1 and the maximum is 7. The higher the overall score, the more severe the symptoms.
  units on a scale | 2.8 [2 to 4]
Baseline Celiac Disease Adherence Test [Median (Full Range); unit: units on a scale] — Celiac Dietary Adherence Test:scores range from 5 to 35, with greater scores indicating poorer adherence;
  units on a scale | 13 [7 to 16]
Baseline IgA anti-human tissue transglutaminase assay (tTG-IgA) [Median (Full Range); unit: unit/liter] — IgA anti-human tissue transglutaminase assay (Inova Diagnostics, Inc., San Diego, USA): negative <20, borderline 20-30, positive >30;
  unit/liter | 12 [2 to 27]
Baseline Fecal elastase-1 levels [Count of Participants; unit: Participants] — Normal range of fecal elastase-1 (Joli Diagnostics, Inc., Buffalo, USA): 200-500 µg/g stool,<200 µg/g stool indicates positive fecal elastase-1 test.
  Participants
    <200 µg/g | 1
    200-500 µg/g | 5
    >500 µg/g | 6

OUTCOME MEASURES:

1. Primary Outcome: Change of Gastrointestinal Symptoms
Description: The average per individual subject on-treatment score in the Celiac Disease Gastrointestinal Symptom Rating Scale (CeD GSRS) domains of Diarrhea, Indigestion, and Abdominal pain comparing active treatment to placebo (i.e. a paired comparison of CeD GSRS on treatment versus on placebo for each subject).
  CeD-GSRS: Each individual sub-section of the 15 sub-sections scores from 1 to 7, with greater scores indicating worse symptoms. A total score can range from 15 -105. This is then divided by 15 to obtain the minimum overall CeD-GSRS score of 1 and maximum of 7. It has 3 domains- Abdominal pain, Indigestion and Diarrhea domains, each domain having a score ranging from 1-7. The higher the overall score, the more severe the symptoms.
Time Frame: Measured at end of each 10- day treatment period
Population: All participants who completed entire study duration were included in the analysis. A comparison of the within-pair differences (delta) in symptom scores after Pancreatic Enzyme Supplement and Placebo treatment, by the Wilcoxon signed rank test.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo Treatment: Participants ingested placebo tablets 6 times daily (with meals and 3 snacks) for 10 days. To facilitate duodenal digestion Omeprazole (20 mg/QD) was co-administered
- PES Treatment: PES treatment was taken 6 times daily with gluten-free meals and 3 snacks. To facilitate duodenal digestion Omeprazole (20 mg/QD) was co-administered.
- Within Participant Difference in Scores Between Treatment Periods: We calculated a delta change between the GSRS scores at end of Placebo treatment and end of PES treatment
Arm/Group | Placebo Treatment | PES Treatment | Within Participant Difference in Scores Between Treatment Periods
Number analyzed (Participants) | 12 | 12 | 12
units on a scale
  GSRS score | 35.75 (12.11) | 37.5 (13.38) | -1.75 (5.83)
  GSRS score: Abdominal pain | 2.5 (1.16) | 2.42 (1.16) | 0.08 (0.79)
  GSRS score: Diarrhea score | 1.25 (0.45) | 1.58 (0.90) | -0.33 (0.65)
  GSRS score: Indigestion score | 2.45 (2.07) | 2.5 (2.07) | -0.18 (2.04)
Statistical Analysis 1: Comparison: Placebo Treatment vs PES Treatment; Test type: Superiority; p = 0.271, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Correlation of Baseline Fecal Elastase and Celiac Disease Gastrointestinal Symptom Response at End of PES Treatment
Description: Baseline fecal elastase measurement will be correlated with Celiac Disease Gastrointestinal Symptom Rating Scale (CeD-GSRS) scores at the end of PES treatment period.
  Celiac Disease Gastrointestinal Symptom Response Scale:scores range from 1 to 7, with greater scores indicating worse symptoms. The minimum score obtainable is 15 and the maximum score obtainable is 105. This is then divided by 15 to obtain the minimum overall CeD-GSRS score of 1 and maximum of 7. It has 3 domains- Abdominal pain, Indigestion and Diarrhea domains, each domain having a score ranging from 1-7. The higher the overall score, the more severe the symptoms.
Time Frame: Baseline visit (fecal elastase levels measured) and end of PES treatment period (CeD-GSRS scores measured)
Population: At the baseline visit, all subjects had their fecal elastase measured from a baseline stool sample. This fecal elastase level was then correlated at the end of the study with a participant's response to treatment. PES treatment response was measured by GSRS scores at the end of PES treatment period.
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Groups:
- Total Participants: Correlation between Baseline fecal elastase measurement and Celiac Disease Gastrointestinal Symptom Rating Scale (CeD-GSRS) scores at the end of PES treatment period.
Arm/Group | Total Participants
Number analyzed (Participants) | 12
Correlation coefficient | 0.223 [-0.198 to 0.646]
Statistical Analysis 1: Comparison: Total Participants; Test type: Other — In order to calculate a correlation between baseline fecal elastase-1 and total CeD-GSRS score on PES treatment vs. placebo treatment, we calculated a Spearman's rank correlation coefficient between the two independent variables; p = 0.995, Spearman rank coefficient

3. Secondary Outcome: Change in Celiac Symptom Index Scores
Description: The average per individual subject on-treatment scores in the Celiac Symptom Index (CSI) comparing PES treatment to placebo.
  For the Celiac Symptom Index: scores range from 16 to 80, with greater scores indicating worse symptoms
  Leffler DA, Dennis M, Edwards George J, Jamma S, Cook EF, Schuppan D, Kelly CP. A validated disease-specific symptom index for adults with celiac disease. Clin Gastroenterol Hepatol. 2009;7:1328-34. PubMed PMID: 19665584.
Time Frame: Measured at the end of each 10-day treatment period
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo Treatment: Evaluated CSI score across all participants during the Placebo treatment
- PES Treatment: Evaluated CSI score across all participants during the PES treatment
- Within Participant Difference in Scores Between Treatment Periods: We calculated a delta change between the CSI scores at the end of Placebo treatment and end of PES treatment.
Arm/Group | Placebo Treatment | PES Treatment | Within Participant Difference in Scores Between Treatment Periods
Number analyzed (Participants) | 12 | 12 | 12
score on a scale | 36.75 (11.62) | 35.92 (9.55) | 0.83 (4.67)
Statistical Analysis 1: Comparison: Placebo Treatment; Test type: Other — In order to evaluate the estimated difference of the effect of Pancreatic Enzyme Supplement versus Placebo for the Celiac Symptom Index (CSI) scores, we used a linear mixed effects model with the nlme package; p = 0.08, Linear Mixed Effects model

ADVERSE EVENTS:
Time Frame: Patients were followed for 34 days which was the entire duration of the study.
Description: Anticipated and unanticipated deaths, serious adverse events, and other adverse events due to any cause, whether related or unrelated to treatment
Groups:
- PES Treatment: Participants ingested PES tablets 6 times daily (with meals and 3 snacks) for 10 days. To facilitate duodenal digestion Omeprazole (20 mg/QD) was co-administered.
Arm/Group | Placebo Treatment | PES Treatment
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
Early termination by the sponsor leading to a small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT02475369/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT02475369/ICF_001.pdf